CLINICAL TRIAL: NCT00861133
Title: Long-Term Cardiac Monitoring for Detection of Atrial Fibrillation After Cryptogenic Stroke
Brief Title: Cryptogenic Stroke Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Transoma Medical (Industry)
Responsible Party: Wim Stegink, Tranoma Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP-008
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2009-05-05 (Estimated); Status verified 2009-05

CONDITIONS: Cryptogenic Stroke
Keywords: cardiac monitor; loop recorder; stroke; ECG; Implantable Loop Recorder; cryptogenic; ILR
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Sleuth AT Implantable ECG Monitoring System — The study device provides monitoring only. It cannot provide intervention or treatment.

SUMMARY:
The purpose of this study is to determine whether the Sleuth Implantable Loop Recorder will enhance detection of latent atrial fibrillation in patients after cryptogenic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Recent stroke (within 30 days) as defined by who has a sudden onset of focal neurological deficits presumed vascular etiology and lasting more than 24 hours.
* Negative brain image for hemorrhagic stroke
* In sinus rhythm at time of enrollment

Exclusion Criteria:

* Know history of atrial fibrillation
* Previous implanted cardiac device (ppM or ICD)
* Serious illness making it unlikely to survive one year
* Known secondary cause of stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-03; Primary Completion 2011-04 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation at one year from Sleuth implantation. | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Krahn, MD, Principal Investigator — Western University, Canada
Locations (1):
- The Ohio State University, Columbus, Ohio, United States